CLINICAL TRIAL: NCT07216937
Title: Effectiveness Comparison of 3D-Printed and Conventional Ear Tip Comfort in Individuals With Hearing in the Normal Range
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Bryan Wong, Assistant Professor of Practice, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00005737
Record Dates: First submitted 2025-10-10; First posted 2025-10-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hearing Aids; 3D Printing
Keywords: hearing aids; 3D printing; hearing healthcare accessibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- In-house Study group_Resin (Experimental): ear tips fabricated using biocompatible resin
  Interventions: Device: BTE hearing aid with compatible earmolds
- Third-party control (Active Comparator): ear tips fabricated by third party manufacturer using biocompatible resin
  Interventions: Device: BTE hearing aid with compatible earmolds
- In-house Study group_FlexibleResin (Experimental): ear tips fabricated using biocompatible flexible resin
  Interventions: Device: BTE hearing aid with compatible earmolds

INTERVENTIONS:
Device: BTE hearing aid with compatible earmolds — Hearing aids will be fit with three different types of customized ear tips. They will only wear each ear tip group for the duration of the test (total = 20 minutes). Hearing aids will be programmed to a simulated mild, flat, sensorineural hearing loss of 40 dB HL from 250-8000Hz. A short washout period will follow completion of testing with ear ear tip group.

SUMMARY:
Access to affordable and timely hearing healthcare remains a major challenge for many individuals, partly due to the high cost and long turnaround time. This study will explore whether 3D-printed ear tips perform as well as or better than standard ear tips in terms of sound quality, comfort, and fit. It will also compare how long each method takes to make and how much each costs.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing thresholds (<25 dB HL) at octave frequencies from 250-8000Hz.
* Normal otoscopy: patent ear canals with normal appearing eardrums and aerated middle ear, bilaterally.
* English speaking.

Exclusion Criteria:

* history of extensive or current outer or middle ear pathology.
* history of extensive outer or middle ear surgery.
* history of neurological or cognitive disorder.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Real Ear Measures | 2nd listening session appointment (15 minutes)
  Evaluation of ear canal acoustics with participant wearing a hearing aid and eartip type (3d party control, in-house_Resin, in-house_FlexResin). Then, a thin microphone tube is placed in the ear canal to measure the average amount gain (dB SPL) across various frequencies (250-8000Hz) while the participant sits in front of a speaker playing sound samples. Results are recorded in gain (dB SPL) across frequencies. Once complete, the eartip type is changed and recording is repeated until all eartip material types have been tested for each individual.
Outer EAR comfort questionnaire | 2nd listening session appointment (10 minutes)
  A validated questionnaire, Outer EAR, will be used to elicit patient perception of physical comfort, acoustic comfort, quality of voice, and overall self-perceived satisfaction. Includes 6 items (5 levels) , with 5 representing best possible function/rating.

SECONDARY OUTCOMES:
Cost | Prior to second listening session appointment (15 minutes)
  The total raw cost ($, dollars US)
Time | Prior to second listening appointment (15 minutes)
  time-to-subject for each eartip type

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona Hearing Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No